CLINICAL TRIAL: NCT06892041
Title: Development of RPBM for Quantitative Assessment of Myofascial Pain
Brief Title: Diffusion MRI for Quantitative Assessment of Myofascial Pain
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 24-07027694; R61AT012270 (NIH)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Masticatory Myofascial Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal: Subjects without masticatory myofascial pain syndrome
- Latent/Active Pain Stage: Subjects with latent or active masticatory myofascial pain syndrome

SUMMARY:
The purpose of this study is to assess the diagnostic accuracy of diffusion MRI for evaluation of the jaw muscles for patients with masticatory myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age
* Ability to give informed consent
* Symptoms meeting criteria for normal or latent/active temporomandibular myofascial pain

Exclusion Criteria:

* Contraindications to MRI scanning including severe obesity or difficulty in laying in a supine position, intracranial clips, metal implants, external metallic devices/objects/clips within 10mm of the head, suspected or confirmed metal in the eyes (history of welding or similar activity), claustrophobia, cardiac pacemaker or pacing wires
* Pregnancy or breast feeding
* Traumatic injury of masticatory muscles or temporomandibular joint within last 12 months
* Mandibular fracture within last 12 months
* Initiation of additional treatment of myofascial pain within the past 1 month
* Received masseter Botox within the last 4 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from the community
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in mean diffusion MRI parameters of temporalis and masseter muscles between patients at the normal stage and those at the latent/active pain stage. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gene Kim, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York University, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Time Frame: Immediately following publication for a minimum of 2 years after completion of the research project
Access Criteria: Anyone who wishes to access the data